CLINICAL TRIAL: NCT03057795
Title: A Phase 2 Study of Nivolumab and Brentuximab Vedotin Consolidation After Autologous Stem Cell Transplantation in Patients With High-Risk Classical Hodgkin Lymphoma
Brief Title: Nivolumab & Brentuximab Vedotin Consolidation After Autologous SCT in Patients With High-Risk Classical Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16378; NCI-2017-00222 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16378 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2017-02-14; First posted 2017-02-20 (Actual); Results first posted 2023-03-23 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Classic Hodgkin Lymphoma; Recurrent Hodgkin Lymphoma; Refractory Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (brentuximab vedotin, nivolumab) (Experimental): Beginning 30-60 days post-ASCT, patients receive brentuximab vedotin IV over 30 minutes and nivolumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Brentuximab Vedotin; Other: Laboratory Biomarker Analysis; Biological: Nivolumab

INTERVENTIONS:
Drug: Brentuximab Vedotin — Given IV
  Other Names: ADC SGN-35; Adcetris; Anti-CD30 Antibody-Drug Conjugate SGN-35; Anti-CD30 Monoclonal Antibody-MMAE SGN-35; Anti-CD30 Monoclonal Antibody-Monomethylauristatin E SGN-35; cAC10-vcMMAE; SGN-35
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial studies how well nivolumab and brentuximab vedotin work after stem cell transplant in treating patients with high-risk classical Hodgkin lymphoma that has come back (recurrent) or does not respond to treatment (refractory). Immunotherapy with monoclonal antibodies, such as nivolumab and brentuximab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the efficacy of nivolumab plus brentuximab vedotin consolidation after autologous stem cell transplantation (ASCT) in participants with relapsed/refractory Hodgkin lymphoma (HL), as assessed by 18-month progression-free survival (PFS).

SECONDARY OBJECTIVES:

I. Estimate the overall survival (OS), the cumulative incidence of relapse/progression, the cumulative incidence of non-relapse mortality (TRM) in participants with relapsed/ refractory HL who receive nivolumab plus brentuximab vedotin consolidation after ASCT.

II. Estimate the overall response rate to nivolumab plus brentuximab vedotin therapy in participants with measurable disease after ASCT.

III. Establish the safety and tolerability of nivolumab plus brentuximab vedotin when used as consolidation after ASCT in participants with relapsed/ refractory HL.

EXPLORATORY OBJECTIVES:

I. Evaluate the Lymphoma Response to Immunomodulatory therapy Criteria (LYRIC) definition of indeterminate response to guide the management of patients regarding treatment past progressive disease.

II. Explore the impact of nivolumab plus brentuximab vedotin therapy on immune reconstitution after ASCT.

III. Explore the prognostic impact of and temporal dynamics of minimal residual disease (MRD) in the peripheral blood as assessed by the next-generation sequencing-based ClonoSEQ platform.

IV. Explore the prognostic impact of 9p24.1 abnormalities in tumor tissue assessed by fluorescence in situ hybridization (FISH) on outcomes after ASCT and nivolumab plus brentuximab vedotin post-ASCT consolidation therapy.

V. Explore the relationship between immune cells and Hodgkin and Reed/Sternberg (HRS) in tumor samples by 6-color quantitative spatial image analysis using the Vectra system, and correlate with outcome after ASCT and nivolumab plus brentuximab vedotin post-ASCT consolidation therapy.

VI. Explore whether genetic alterations (e.g. gene expression profiles or genetic mutations) in HL tumor samples are associated with outcome after ASCT and nivolumab plus brentuximab vedotin post-ASCT consolidation therapy.

OUTLINE:

Beginning 30-60 days post-ASCT, patients receive brentuximab vedotin intravenously (IV) over 30 minutes and nivolumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 100 days, at 3, 6, 12, and 18 months from start of treatment, and then biannually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent
* Agreement to allow the use of archival tissue from pre-ASCT tumor biopsies

  * If unavailable, exceptions may be granted with study principal investigator (PI) approval
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Histologically confirmed diagnosis of classical Hodgkin lymphoma (excluding nodular lymphocyte predominant Hodgkin lymphoma) according to the World Health Organization (WHO) classification, with hematopathology review at the participating institution
* Have high-risk relapsed or refractory Hodgkin lymphoma (HL), defined as at least one of the following:

  * Primary refractory disease to front-line therapy
  * Relapse within 1 year of completing front-line therapy
  * Extranodal involvement at the time of pre-ASCT relapse
  * B symptoms at pre-ASCT relapse
  * More than one type of pre-ASCT salvage therapy required
* Planning to receive or have received autologous stem cell transplantation (ACST) per institutional standards as part of standard of care

  * Pre-ASCT participants may consent but will not be eligible to begin treatment until after ASCT, and will have to fulfill all inclusion and exclusion criteria before starting protocol
  * All participants must initiate day 1 of protocol therapy within 30-60 days post stem cell reinfusion; study PI can grant exception for a patient to start as late as 75 days post stem cell reinfusion with a reasonable justification for a delay (e.g. recovery from post -ASCT toxicity) and this will not be a protocol deviation, nor require an exception to be filled
* Recovery from ASCT toxicity as defined as outpatient status, able to drink, eat normally, and do not need intravenous hydration prior to day 1 of therapy
* Achieved at least stable disease to salvage treatment determined by positron emission tomography (PET)/computed tomography (CT) using 2014 Lugano Classification prior to ASCT
* Brentuximab vedotin naive OR had at least stable disease by Lugano Classification to prior brentuximab vedotin treatment
* Absolute neutrophil count (ANC) >= 1000/mm^3
* Platelets >= 50,000/mm^3
* Hemoglobin >= 8 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or 3 x ULN for Gilbert's disease
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN
* Creatinine clearance >= 40 mL/min per 24 hour urine collection or the Cockcroft-Gault formula

  * Calculated per institutional standard
* Forced expiratory volume in one second (FEV1) and carbon monoxide diffusion capacity (DLCO) (adjusted for hemoglobin [Hb]) >= 50% adjusted
* Women of childbearing potential (WOCBP) only: Negative urine or serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG])

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Woman of childbearing potential (WOCBP): use two effective methods of contraception (hormonal or barrier method) or be surgically sterile, or abstain from heterosexual activity for the course of the study through 7 months post last dose of nivolumab

  * WOCBP defined as not being surgically sterilized or have not been free from menses for > 1 year
  * Male: use two effective methods of contraception (barrier method) or abstain from heterosexual activity with the first dose of study therapy through 7 months post last dose of nivolumab

Exclusion Criteria:

* Post-ASCT anti-lymphoma or investigational therapy; immediate post-ASCT consolidative radiation therapy is allowed as long as it occurs prior to initiation of study therapy; baseline imaging and pulmonary function tests (PFTs) must be performed after completion of radiation
* Previous allogeneic transplant
* Total carmustine (BCNU) dose of > 600 mg/m^2 with prior treatments including transplant conditioning regimen
* Live vaccine within 30 days prior to day 1 of protocol therapy (e.g. measles, mumps, rubella, varicella, yellow fever, rabies, Bacillus Calmette-Guerin [BCG], oral polio vaccine, and oral typhoid)
* Refractory to prior brentuximab vedotin (i.e. progression while on treatment)
* Refractory to prior anti-PD-1/PD-L1 agent
* History of prior >= grade 3 hypersensitivity to either brentuximab vedotin or nivolumab
* History of another primary malignancy that has not been in remission for at least 3 years; exceptions include:

  * Basal cell carcinoma of the skin or
  * Squamous cell carcinoma of the skin that has undergone potentially curative therapy or
  * In situ cervical cancer
* Known active central nervous system (CNS) involvement by lymphoma, including parenchymal and/or lymphomatous meningitis
* History of progressive multifocal leukoencephalopathy (PML)
* Grade >= 2 peripheral neuropathy at the present time
* Prior diagnosis of inherited or acquired immunodeficiency
* Condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration; exceptions are:

  * Inhaled or topical steroids and
  * Adrenal replacement doses > 10 mg daily prednisone equivalents in the absence of active autoimmune disease
* Uncontrolled illness including ongoing or active infection
* History of or active pneumonitis or interstitial lung disease:

  * For history of pneumonitis to be an exclusion, patient had to have required supplemental oxygen or corticosteroid treatment; radiographic changes alone are not an exclusion
* An active, known or suspected autoimmune disease; the following are exceptions:

  * Vitiligo
  * Hemolytic anemia associated with the lymphoma (history of or at the present time)
  * Type I diabetes mellitus
  * Residual hypothyroidism due to autoimmune condition only requiring hormone replacement
  * Psoriasis not requiring systemic treatment, or
  * Conditions not expected to recur in the absence of an external trigger
* Active or known history (standard pre-ASCT assessments) of:

  * Hepatitis B or C infection
  * Human immunodeficiency virus (HIV)
  * Acquired immunodeficiency syndrome (AIDS)
* Women who are pregnant or lactating
* History of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association Class III-IV within 6 months prior to day 1 of protocol therapy
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2026-03-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Herrera, Principal Investigator — City of Hope Medical Center
Locations (6):
- United States (6):
  - City of Hope Medical Center, Duarte, California
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - M D Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Herrera AF, Chen L, Nieto Y, Holmberg L, Johnston P, Mei M, Popplewell L, Armenian S, Cao T, Farol L, Sahebi F, Spielberger R, Chen R, Nademanee A, Puverel S, Nwangwu M, Lee P, Song J, Skarbnik A, Kennedy N, Peters L, Rosen ST, Kwak LW, Forman SJ, Feldman T. Brentuximab vedotin plus nivolumab after autologous haematopoietic stem-cell transplantation for adult patients with high-risk classic Hodgkin lymphoma: a multicentre, phase 2 trial. Lancet Haematol. 2023 Jan;10(1):e14-e23. doi: 10.1016/S2352-3026(22)00318-0. Epub 2022 Nov 17. PMID 36403579

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three subjects consented but did not participate in the study. Two subjects withdrew consent and one subject became ineligible due to developmental of interstitial pneumonia after consent before screening.
Groups:
- Brentuximab Vedotin 1.8 mg/kg + Nivolumab 3 mg/kg Q21 Days: Beginning 30-60 days post-ASCT, patients receive brentuximab vedotin IV over 30 minutes and nivolumab IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Brentuximab Vedotin: Given IV Nivolumab: Given IV
Period: Overall Study
Arm/Group | Brentuximab Vedotin 1.8 mg/kg + Nivolumab 3 mg/kg Q21 Days
Started | 59
Completed | 59
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects were screened, enrolled, and treated with brentuximab vedotin plus nivolumab.
Arm/Group | Brentuximab Vedotin 1.8 mg/kg + Nivolumab 3 mg/kg Q21 Days
Number analyzed (Participants) | 59
Age, Continuous [Median (Full Range); unit: years] | 30 [23 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 18 Months
Description: Progression-free survival will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error. When there is no censoring in progression-free survival prior to 18 months after the first dose of study treatment, the observed 18-month progression-free survival will be compared to the baseline of 65% by one-sided exact test of binomial proportion. In case of censoring in progression-free survival prior to 18 months after the first dose of study treatment, the Kaplan-Meier estimate for 18-month progression-free survival along with the Greenwood standard error estimator will be used for the testing of null hypothesis at 65%. Hodgkin Lymphoma(HL) response/progression was evaluated using 2014 Lugano Classification [Cheson, Journal of Clinical Oncology 2014 Sep 20;32(27):3059-68].
Time Frame: From the first dose of study treatment to the first observation of disease relapse/progression or death from any cause, whichever occurs first, assessed at 18 months.
Measure: Number (95% Confidence Interval); unit: percentage of survival probability
Arm/Group | Brentuximab Vedotin 1.8 mg/kg + Nivolumab 3 mg/kg Q21 Days
Number analyzed (Participants) | 59
percentage of survival probability | 94 [84 to 98]

2. Secondary Outcome: Overall Survival at 18 Months
Description: Overall survival will be estimated using the product-limit method of Kaplan and Meier along with the Greenwood estimator of standard error.
Time Frame: From the first dose of study treatment to death from any cause, assessed up to 18 months
Measure: Number (95% Confidence Interval); unit: percentage of survival probability
Arm/Group | Brentuximab Vedotin 1.8 mg/kg + Nivolumab 3 mg/kg Q21 Days
Number analyzed (Participants) | 59
percentage of survival probability | 98 [88 to 100]

ADVERSE EVENTS:
Time Frame: From the date of the first dose up to 48 months.
Arm/Group | Brentuximab Vedotin 1.8 mg/kg + Nivolumab 3 mg/kg Q21 Days
All-Cause Mortality (participants affected / at risk) | 1/59
Serious Adverse Events (participants affected / at risk) | 19/59
Other Adverse Events (participants affected / at risk) | 59/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brentuximab Vedotin 1.8 mg/kg + Nivolumab 3 mg/kg Q21 Days (N=59)
Cardiac arrest (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 8 (9)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Eggerthella lenta pneumonia (Infections and infestations) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastric Neuroendocrine Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brentuximab Vedotin 1.8 mg/kg + Nivolumab 3 mg/kg Q21 Days (N=59)
ANEMIA (Blood and lymphatic system disorders) | 11 (25)
ASYMPTOMATIC CT SCAN CHANGES (Cardiac disorders) | 1 (6)
PALPITATIONS (Cardiac disorders) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 6 (9)
SINUS TACHYCARDIA (Cardiac disorders) | 21 (33)
MILD IMBALANCE (Ear and labyrinth disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 5 (11)
INCREASED TSH (Endocrine disorders) | 1 (1)
BLURRED VISION (Eye disorders) | 2 (2)
EYE PAIN (Eye disorders) | 1 (1)
SCLERAL DISORDER (Eye disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 (19)
BLOATING (Gastrointestinal disorders) | 2 (2)
COLITIS (Gastrointestinal disorders) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 6 (9)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 18 (26)
DIVERTICULITIS (Gastrointestinal disorders) | 1 (1)
DRY MOUTH (Gastrointestinal disorders) | 4 (4)
DYSPEPSIA (Gastrointestinal disorders) | 6 (6)
DYSPHAGIA (Gastrointestinal disorders) | 2 (2)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (3)
ILEUS (Gastrointestinal disorders) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 2 (3)
NAUSEA (Gastrointestinal disorders) | 19 (23)
ORAL PAIN (Gastrointestinal disorders) | 2 (2)
ORAL THRUSH (Gastrointestinal disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 13 (14)
CHILLS (General disorders) | 15 (19)
EDEMA LIMBS (General disorders) | 1 (1)
FATIGUE (General disorders) | 27 (40)
FEVER (General disorders) | 14 (18)
FLU LIKE SYMPTOMS (General disorders) | 5 (6)
IMBALANCE (General disorders) | 1 (1)
INFUSION RELATED REACTION (General disorders) | 4 (6)
INJECTION SITE REACTION (General disorders) | 2 (2)
MALAISE (General disorders) | 4 (4)
NONCARDIAC CHEST PAIN (General disorders) | 4 (4)
PAIN (General disorders) | 6 (7)
VOD (IMMUNE RELATED) (Hepatobiliary disorders) | 1 (1)
ALLERGIC REACTION (Immune system disorders) | 2 (2)
CDIFF (Infections and infestations) | 1 (1)
HEPATITIS VIRAL (Infections and infestations) | 1 (1)
LARYNGITIS (Infections and infestations) | 1 (1)
LUNG INFECTION (Infections and infestations) | 2 (2)
MYCOBACTERIUM AVIUM INTRACELLULARE (Infections and infestations) | 1 (1)
PHARYNGITIS (Infections and infestations) | 1 (1)
RHINITIS INFECTIVE (Infections and infestations) | 1 (1)
RHINOVIRUS UPPER RESPIRATORY (Infections and infestations) | 1 (1)
SKIN INFECTION (Infections and infestations) | 2 (2)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 25 (39)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2)
VAGINAL INFECTION (Infections and infestations) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 1 (1)
BRUISING (Injury, poisoning and procedural complications) | 1 (1)
DOG BITE (Injury, poisoning and procedural complications) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (3)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 14 (22)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 2 (3)
AMYLASE DECREASED (Investigations) | 1 (4)
APPETITE (Investigations) | 1 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 16 (22)
BASOPHILS COUNT INCREASED (Investigations) | 1 (3)
BLAST COUNT INCREASED (Investigations) | 1 (2)
BLOOD BILIRUBIN INCREASED (Investigations) | 5 (7)
BUN INCREASED (Investigations) | 1 (1)
CARBON DIOXIDE ELEVATED (Investigations) | 1 (3)
CARDIAC TROPONIN I INCREASED (Investigations) | 1 (1)
CHLORIDE INCREASED (Investigations) | 1 (2)
CHOLESTEROL HIGH (Investigations) | 1 (2)
CREATININE INCREASED (Investigations) | 4 (7)
EOSINOPHIL COUNT INCREASED (Investigations) | 1 (1)
EOSINOPHILS COUNT INCREASED (Investigations) | 1 (2)
ERYTHROCYTE SEDRATE ELEVATED (Investigations) | 1 (1)
FORCED EXPIRATORY VOLUME DECREASED (Investigations) | 1 (1)
HYPERLIPIDEMIA (Investigations) | 1 (8)
INCREASE IN STOOL FREQUENCY (Investigations) | 1 (1)
LACTOSE DEHYDROGENASE INCREASED (Investigations) | 7 (14)
LIPASE INCREASED (Investigations) | 3 (4)
LYMPHOCYTE COUNT DECREASED (Investigations) | 14 (44)
NEUTROPHIL COUNT DECREASED (Investigations) | 25 (49)
NEUTROPHIL COUNT INCREASED (Investigations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 8 (14)
SATIETY (Investigations) | 1 (2)
SERUM AMYLASE INCREASED (Investigations) | 2 (3)
SKIN NODULE (Investigations) | 1 (1)
URIC ACID DECREASED (Investigations) | 2 (4)
WEIGHT GAIN (Investigations) | 6 (8)
WEIGHT LOSS (Investigations) | 13 (26)
WHITE BLOOD CELL DECREASED (Investigations) | 16 (36)
ANOREXIA (Metabolism and nutrition disorders) | 6 (6)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPERNATREMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPERURICEMIA (Metabolism and nutrition disorders) | 4 (9)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 4 (6)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 3 (4)
HYPOKALEMIA (Metabolism and nutrition disorders) | 3 (5)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (2)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 4 (4)
OBESITY (Metabolism and nutrition disorders) | 4 (5)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 15 (19)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 7 (7)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 4 (4)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 13 (20)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 (3)
DIZZINESS (Nervous system disorders) | 3 (4)
DYSESTHESIA (Nervous system disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 11 (14)
PARESTHESIA (Nervous system disorders) | 2 (2)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 11 (27)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 31 (46)
PRESYNCOPE (Nervous system disorders) | 1 (1)
SYNCOPE (Nervous system disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 9 (14)
DEPRESSION (Psychiatric disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 7 (9)
RESTLESSNESS (Psychiatric disorders) | 1 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 (2)
DYSURIA (Renal and urinary disorders) | 2 (2)
HEMATURIA (Renal and urinary disorders) | 3 (3)
PROTEINURIA (Renal and urinary disorders) | 3 (3)
URINE DISCOLORATION (Renal and urinary disorders) | 2 (2)
DYSPAREUNIA (Reproductive system and breast disorders) | 1 (1)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1)
PREMATURE MENOPAUSE (Reproductive system and breast disorders) | 1 (1)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 2 (2)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 1 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 23 (28)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 16 (21)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 2 (4)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3 (4)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 9 (9)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 7 (17)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 (2)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 7 (8)
STREP THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DOG BITE (Skin and subcutaneous tissue disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 (5)
ERYTHRODERMA (Skin and subcutaneous tissue disorders) | 1 (1)
FACIAL ACNE (Skin and subcutaneous tissue disorders) | 1 (2)
HEAT RASH (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 5 (5)
PALMARPLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 1 (1)
PLANTAR WART (Skin and subcutaneous tissue disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 10 (12)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 (2)
RASH MACULOPAPULAR (Skin and subcutaneous tissue disorders) | 17 (27)
RASH/OISON IVY (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN INDURATION (Skin and subcutaneous tissue disorders) | 1 (1)
SMALL LESION ON LEFT THIGH (Skin and subcutaneous tissue disorders) | 1 (1)
HOT FLASHES (Vascular disorders) | 3 (3)
HYPERTENSION (Vascular disorders) | 25 (54)
HYPOTENSION (Vascular disorders) | 15 (23)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT03057795/Prot_SAP_000.pdf